CLINICAL TRIAL: NCT02792946
Title: Compare the Efficacy and Safety of Surfolase CR Tablet With Surfolase Capsule in Patients With Acute Bronchitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hyundai Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HT-002-05
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2016-06

CONDITIONS: Acute Bronchitis
MeSH Terms: conditions — Bronchitis | interventions — ambroxol-theophylline-7-acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sulfolase CR (200mg, QD) (Experimental): for 7 days with or without meal
  Interventions: Drug: Acebrophylline
- Sulfolase Capsule (100mg, BID) (Active Comparator): for 7 days with or without meal
  Interventions: Drug: Acebrophylline

INTERVENTIONS:
Drug: Acebrophylline

SUMMARY:
Compare the efficacy and safety of surfolase CR tablet with surfolate capsule in patients with acute bronchitis

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 19 to 65 years, inclusive
2. Patients with acute bronchitis which is accompanied with a cough which includes sputum within 48 hours and has over 5 for Bronchitis severity score (BSS) at Screening
3. Patients who agreed to participate clinical trial and sign on informed consent form

Exclusion Criteria:

1. Patients who are suspicious or diagnosed for pneumonia
2. Patients with chronic bronchitis, Chronic Obstructive Pulmonary Disease (COPD), bronchiolitis, asthma, bronchial asthma
3. Patients with active infection who needs administration of antibiotics
4. Patients with myocardial infarction, congestive heart failure
5. Patients with renal disorder or liver disorder
6. Patients with hypotension or hypertension
7. Patients with history of epilepsy
8. Patients with hyperthyroidism
9. Patients with gastroduodenal ulcer
10. Patients with sever hypoxemia
11. Patients who are in drug or therapy or planned to have;

    * antibiotics, anti-virus, angiotensin converting enzyme (ACE) inhibitor and systemic or inhalation glucocorticosteroids: from 2 weeks prior to administration of investigational product to termination of clinical trial
    * Angiotension II receptor blocker (ARB), secretolytics/mucolytics, expectorants, antitussives, a herb medicines which has antitussive or expectorant effect: from 2 days prior to administration of investigational product to termination of clinical trial
    * Analgesics except acetaminophen, antihistamines, β2-agonists, bronchodilators which includes anticholinergic agents, xanthine derivatives, central nervous system stimulants, drug which is known for interaction between acebrophylline (cimetidine, alloprinol, oral anticoagulants, furosemide, reserpine, barbiturates, phenytoin) and symtomatic therapy for other therapy for acute bronchitis: whole period for clinical trial
12. Smokers
13. Patients who has history for drug hypersensitivity or allergic reaction in component of investigational product or similar drug
14. Patients with pregnant and/or have breast feeding.
15. Patients with no intention to use appropriate contraceptives or has a plan to become pregnant
16. Patients who had an administrationb of other investigational product or medical device for clinical trial 4 weeks prior to participation of clinical trial
17. Patients who are identified as inappropriate by other investigators to participate clinical trial

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in baseline to Day 7 for total number of Bronchitis Severity Score (BSS) | Baseline, At Day 7

SECONDARY OUTCOMES:
Change from Baseline in baseline to Day 7 for number of BSS per symptom | Baseline, At Day 7
Response rate at Day 7 | Baseline, At Day 7

IPD SHARING:
Plan to Share IPD: No